CLINICAL TRIAL: NCT01146834
Title: A Prospective Randomized Trial Comparing Three Different Peripheral Stem Cell Mobilization Regimens in Patients With Symptomatic Multiple Myeloma or Lymphoma
Brief Title: Trial of Three Stem Cell Mobilization Regimens for Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1005011049; X05324 (Other Grant/Funding Number: Millennium)
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Filgrastim; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF (Experimental): VELCADE at 1.3 mg/m2 IVP on days 1, 4, 8 and 11 in combination with high-dose cyclophosphamide at 2.0 g/m2 on day 4. G-CSF is given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day. Pheresis will commence once ANC of 1.5 is reached.
  Interventions: Drug: bortezomib (Velcade); Drug: cyclophosphamide; Drug: G-CSF
- Arm B: VELCADE & G-CSF (Experimental): VELCADE at 1.3 mg/m2 IVP on days 1, 4, 8 and 11. G-CSF is given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day. Day 12 start pheresis collection
  Interventions: Drug: bortezomib (Velcade); Drug: G-CSF
- Arm C: CYCLOPHOSPHAMIDE & G-CSF (Experimental): High-dose cyclophosphamide at 2.0 g/m2 on day 1. G-CSF is given for ten (+/- two) consecutive days starting on day 2 at a dose of 10 micrograms/kg/day. Pheresis will commence once ANC of 1.5 is reached.
  Interventions: Drug: cyclophosphamide; Drug: G-CSF
- Arm D: PLERIXAFOR & G-CSF (Experimental): G-CSF is given for ten (+/- two) consecutive days starting on day 1 at a dose of 10 micrograms/kg/day. Plerixafor is given on day 4, approximately 11 hours prior to stem cell collection attempt on Day 5. Both G-CSF and plerixafor are continued daily until collection is complete. Pheresis will commence for everyone on Day 5 regardless of ANC status.
  Interventions: Drug: G-CSF; Drug: Plerixafor
- Arm E: PLERIXAFOR, VELCADE, & G-CSF (Experimental): Bortezomib at 1.3 mg/m2 IVP on days 1, 4, 8 and 11. G-CSF is given for ten (+/- wo) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day.
  Plerixafor is given on day 12, approximately 11 hours prior to stem cell collection attempt and is continued daily until collection is complete. Pheresis will commence for everyone on Day 13 regardless of ANC status.
  Interventions: Drug: bortezomib (Velcade); Drug: G-CSF; Drug: Plerixafor

INTERVENTIONS:
Drug: bortezomib (Velcade) — 1.3 mg/m2 IVP on days 1, 4, 8 and 11
  Other Names: Velcade
  Arms: Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF; Arm B: VELCADE & G-CSF; Arm E: PLERIXAFOR, VELCADE, & G-CSF
Drug: cyclophosphamide — 2.0 g/m2 (day 4 for Arm A and day 1 for Arm C)
  Other Names: Cytoxan
  Arms: Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF; Arm C: CYCLOPHOSPHAMIDE & G-CSF
Drug: G-CSF — given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day (start on day 2 for Arm C and start on Day 1 for Arm D)
  Other Names: Filgrastim; Neupogen
Drug: Plerixafor — plerixafor is given on day 4, approximately 11 hours prior to stem cell collection attempt on Day 5, plerixafor daily until stem cell collection is complete (Arm D), start on Day 12, approximately 11 hours prior to stem cell collection attempt and plerixafor daily until collection if complete (Arm E)
  Other Names: Mozobil
  Arms: Arm D: PLERIXAFOR & G-CSF; Arm E: PLERIXAFOR, VELCADE, & G-CSF

SUMMARY:
This phase III randomized trial compares three different peripheral stem cell mobilization regimens for patients with multiple myeloma who have received primary induction therapy or other therapies. Up to 180 patients will be enrolled. Patients eligible for treatment will be randomized to one of the three following mobilization regimens:

Arm A = VELCADE, CYCLOPHOSPHAMIDE, & G-CSF Arm B = VELCADE & G-CSF Arm C = CYCLOPHOSPHAMIDE & G-CSF Arm D = PLERIXAFOR & G-CSF Arm E = PLERIXAFOR, VELCADE, & G-CSF

DETAILED DESCRIPTION:
PRIMARY STUDY OBJECTIVES

• To compare the efficacy of the following peripheral stem cell mobilization regimens for MM: i. High dose cyclophosphamide, VELCADE, and G-CSF ii. VELCADE and G-CSF iii. High dose cyclophosphamide and G-CSF

SECONDARY STUDY OBJECTIVES

• To evaluate biomarkers as surrogate markers of mobilization in each arm To evaluate changes in tumor mass as defined by standard response parameters. To evaluate the safety of each of the arms.

This phase III randomized trial compares three different peripheral stem cell mobilization regimens for patients with multiple myeloma who have received primary induction therapy

Primary Endpoints

a) Percentage of patients able to collect >6 x 106 CD34+ cells/kg in < 2 collections.

Secondary Endpoints

1. Engrafting: Neutrophil recovery (ANC >0.5 of <12 days), Plt recovery (>20K untransfused <20 days)) after mel 200 based transplant.
2. Toxicities

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Confirmed diagnosis of multiple myeloma
* Age > than 18 years at the time of signing the informed consent form.
* Karnofsky performance status above 60%
* Patients must be within 30 days of completing induction therapy.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control .
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Life expectancy > 12 weeks.
* Subjects must have a MUGA scan or echo with LVEF >50%
* Subjects must meet the following laboratory parameters:

  1. Absolute neutrophil count (ANC) ≥1500 cells/mm3
  2. Platelets count ≥ 50,000/mm3
  3. Hemoglobin > 9.0 g/dL
  4. Serum SGOT/AST <3.0 x upper limits of normal (ULN)
  5. Serum SGPT/ALT <3.0 x upper limits of normal (ULN)
  6. Serum creatinine < 2.5 mg/dL or creatinine clearance > 40ml/min
  7. Serum total bilirubin < 1.5 x ULN

Exclusion Criteria:

* Patients with (no measurable monoclonal protein, free light chains, and/or M-spike in blood or urine) unless measurable disease is available with imaging techniques such as MRI and PET scan.
* History of allergic reactions to compounds containing boron, mannitol, VELCADE
* Prior history of other malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless disease free for > = 5 years.
* NYHA Class III or IV heart disease. History of active unstable angina, congestive heart disease, severe uncontrolled cardiac arrhythmia, electrocardiographic evidence of acute ischemia, active conduction system abnormalities or myocardial infarction within 6 months prior to enrollment. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Female patients who are pregnant or breastfeeding. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Known HIV or hepatitis A, B, or C positivity---ONLY IF ACTIVE
* Active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Any concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place him/her at unacceptable risk
* Patient has > = Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has received other investigational drugs with 14 days before enrollment
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (5):
- United States (5):
  - Emory University, Atlanta, Georgia
  - New York University Cancer Institute, New York, New York
  - Columbia Presbyterian Medical Center):, New York, New York
  - Memorial Sloan-Kettering Cancer Center):, New York, New York
  - Weill Cornell Medical College, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF: VELCADE at 1.3 mg/m2 IVP on days 1, 4, 8 and 11 in combination with high-dose cyclophosphamide at 2.0 g/m2 on day 4. G-CSF is given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day. Pheresis will commence once ANC of 1.5 is reached.
  bortezomib (Velcade): 1.3 mg/m2 IVP on days 1, 4, 8 and 11
  cyclophosphamide: 2.0 g/m2 (day 4 for Arm A and day 1 for Arm C)
  G-CSF: given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day (start on day 2 for Arm C)
- Arm B: VELCADE & G-CSF: VELCADE at 1.3 mg/m2 IVP on days 1, 4, 8 and 11. G-CSF is given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day. Day 12 start pheresis collection
  bortezomib (Velcade): 1.3 mg/m2 IVP on days 1, 4, 8 and 11
  G-CSF: given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day (start on day 2 for Arm C)
- Arm C: CYCLOPHOSPHAMIDE & G-CSF: High-dose cyclophosphamide at 2.0 g/m2 on day 1. G-CSF is given for ten (+/- two) consecutive days starting on day 2 at a dose of 10 micrograms/kg/day. Pheresis will commence once ANC of 1.5 is reached.
  cyclophosphamide: 2.0 g/m2 (day 4 for Arm A and day 1 for Arm C)
  G-CSF: given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day (start on day 2 for Arm C)
- Arm E: PLERIXAFOR, VELCADE, & G-CSF: Bortezomib at 1.3 mg/m2 IVP on days 1, 4, 8 and 11. G-CSF is given for ten (+/- wo) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day.
  Plerixafor is given on day 12, approximately 11 hours prior to stem cell collection attempt and is continued daily until collection is complete. Pheresis will commence for everyone on Day 13 regardless of ANC status.
  bortezomib (Velcade): 1.3 mg/m2 IVP on days 1, 4, 8 and 11
  G-CSF: given for ten (+/- two) consecutive days starting on day 9 at a dose of 10 micrograms/kg/day (start on day 2 for Arm C and start on Day 1 for Arm D)
  Plerixafor: plerixafor is given on day 4, approximately 11 hours prior to stem cell collection attempt on Day 5, plerixafor daily until stem cell collection is complete (Arm D), start on Day 12, approximately 11 hours prior to stem cell collection attempt and plerixafor daily until collection if complete (Arm E)
Period: Overall Study
Arm/Group | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF | Arm B: VELCADE & G-CSF | Arm C: CYCLOPHOSPHAMIDE & G-CSF | Arm D: PLERIXAFOR & G-CSF | Arm E: PLERIXAFOR, VELCADE, & G-CSF
Started | 20 | 4 | 23 | 0 | 0
Completed | 17 | 4 | 21 | 0 | 0
Not Completed | 3 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects enrolled in Arm D and E.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF | Arm B: VELCADE & G-CSF | Arm C: CYCLOPHOSPHAMIDE & G-CSF | Arm D: PLERIXAFOR & G-CSF | Arm E: PLERIXAFOR, VELCADE, & G-CSF | Total
Number analyzed (Participants) | 20 | 4 | 23 | 0 | 0 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  |  | 0
  Between 18 and 65 years | 15 | 4 | 11 |  |  | 30
  >=65 years | 5 | 0 | 12 |  |  | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 5 |  |  | 17
  Male | 10 | 2 | 18 |  |  | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 |  |  | 2
  Not Hispanic or Latino | 19 | 3 | 22 |  |  | 44
  Unknown or Not Reported | 0 | 1 | 0 |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  |  | 0
  Asian | 0 | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  | 0
  Black or African American | 5 | 2 | 8 |  |  | 15
  White | 14 | 1 | 12 |  |  | 27
  More than one race | 0 | 0 | 0 |  |  | 0
  Unknown or Not Reported | 1 | 1 | 3 |  |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Able to Collect >=6 x 106 CD34+ Cells/kg in <= 2 Collections.
Description: The primary endpoint in all five treatment arms is the percentage of patients who are able to achieve greater than 6 x 106 CD34+ stems cells/kg harvested (defined as effectiveness). Note that no patients were enrolled Arm D and Arm E.
Time Frame: 36 months
Population: Arm A: 20 patients were enrolled but only 17 were evaluable. Arm C: 23 patients enrolled but only 21 were evaluable. Arm D and Arm E of the study did not accrue any subjects, therefore the number of participants analyzed for this outcome measure is 0 for both arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF | Arm B: VELCADE & G-CSF | Arm C: CYCLOPHOSPHAMIDE & G-CSF | Arm D: PLERIXAFOR & G-CSF | Arm E: PLERIXAFOR, VELCADE, & G-CSF
Number analyzed (Participants) | 17 | 4 | 21 | 0 | 0
Participants | 11 | 0 | 14 |  |
Statistical Analysis 1: Comparison: Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF vs Arm C: CYCLOPHOSPHAMIDE & G-CSF; Arm B was initially closed due to low accrual, and Arms D and E were also closed due to no accrual. Arms A and C also had very low accrual. Therefore, the comparison of the primary outcome between Arms A and C is for exploratory purposes only; Test type: Superiority; p = 0.90, Chi-squared; Risk Difference (RD) = -0.02, 95% CI 2-sided [-0.32 to 0.28]

2. Secondary Outcome: Number of Patients Who Achieved Neutrophil Recovery After Melphalan 200 Based Transplant
Description: Number of patients who achieved neutrophil recovery after Melphalan 200 based transplant in 20 days or fewer. Neutrophil recovery is defined as an absolute neutrophil count of greater than 0.5 k/uL for three consecutive days.
Time Frame: 20 days post-transplant
Population: Data analyzed only for patients who went on to receive a stem cell transplant after mobilization. 25 subject did not receive a stem cell transplant after mobilization and therefore are not included in the analysis. However, no statistical test can be performed because the outcome proportion was 100% in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF | Arm B: VELCADE & G-CSF | Arm C: CYCLOPHOSPHAMIDE & G-CSF | Arm D: PLERIXAFOR & G-CSF | Arm E: PLERIXAFOR, VELCADE, & G-CSF
Number analyzed (Participants) | 7 | 4 | 11 | 0 | 0
Participants | 7 | 4 | 11 | 0 | 0

3. Secondary Outcome: Number of Patients Who Achieved Platelet Recovery After Melphalan 200 Based Transplant
Description: Number of patients who achieved platelet recovery after Melphalan 200 based transplant in 20 days or fewer. Platelet recovery is defined as a platelet count of greater than 20,000, untransfused, for three consecutive days.
Time Frame: 20 days post-transplant
Population: Data analyzed only for patients who went on to receive a stem cell transplant after mobilization. 25 subject did not receive a stem cell transplant after mobilization and therefore are not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF | Arm B: VELCADE & G-CSF | Arm C: CYCLOPHOSPHAMIDE & G-CSF | Arm D: PLERIXAFOR & G-CSF | Arm E: PLERIXAFOR, VELCADE, & G-CSF
Number analyzed (Participants) | 7 | 4 | 11 | 0 | 0
Participants | 4 | 1 | 9 | 0 | 0
Statistical Analysis 1: Comparison: Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF vs Arm C: CYCLOPHOSPHAMIDE & G-CSF; Test type: Superiority; p = 0.25, Fisher Exact; Risk Difference (RD) = -0.25, 95% CI 2-sided [-0.68 to 0.18]

ADVERSE EVENTS:
Time Frame: Patients who do not withdraw consent will be followed for survival after end of treatment on a monthly to bi-monthly basis or until death, whichever occurs first. Patients removed from study for unacceptable adverse events will be followed for life every 6 months, unless they withdraw consent.
Description: Arm D and Arm E did not enrolled any patients
Arm/Group | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF | Arm B: VELCADE & G-CSF | Arm C: CYCLOPHOSPHAMIDE & G-CSF | Arm D: PLERIXAFOR & G-CSF | Arm E: PLERIXAFOR, VELCADE, & G-CSF
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/4 | 0/23 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/4 | 1/23 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 8/20 | 4/4 | 18/23 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF (N=20) | Arm B: VELCADE & G-CSF (N=4) | Arm C: CYCLOPHOSPHAMIDE & G-CSF (N=23) | Arm D: PLERIXAFOR & G-CSF (N=0) | Arm E: PLERIXAFOR, VELCADE, & G-CSF (N=0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: VELCADE, CYCLOPHOSPHAMIDE, & G-CSF (N=20) | Arm B: VELCADE & G-CSF (N=4) | Arm C: CYCLOPHOSPHAMIDE & G-CSF (N=23) | Arm D: PLERIXAFOR & G-CSF (N=0) | Arm E: PLERIXAFOR, VELCADE, & G-CSF (N=0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 4 | 2 | 8 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 8 | 2 | 5 | 0 | 0
Platelet count decreased (Investigations) | 7 | 4 | 11 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 2 | 7 | 0 | 0
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 6 | 0 | 6 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 0
Gallbladder Pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
bone pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Serum creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 0 | 2 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0
bloating (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vulval infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Other, Eye twitch (Eye disorders) | 1 | 0 | 0 | 0 | 0
bruising; extremity (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Arm B: VELCADE & G-CSF was closed to further enrollment due to futility in 2013. Arm C: CYCLOPHOSPHAMIDE & G-CSF was closed in 2015 due to futility. Early termination of Arm B and Arm C will limit the sample size for those treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT01146834/Prot_SAP_000.pdf